CLINICAL TRIAL: NCT02726048
Title: Simplus and Eson Non-Invasive Ventilation (NIV) Evaluation - Germany
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Fisher & Paykel Healthcare placed an administrative hold on the Simplus and Eson Non-Invasive Ventilation Evaluation study being conducted at Charite, Berlin
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA178
Record Dates: First submitted 2016-03-29; First posted 2016-04-01 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Obesity Hypoventilation Syndrome; Obstructive Sleep Apnea; Chronic Obstructive Pulmonary Disease; Neuromuscular Disease
MeSH Terms: conditions — Obesity Hypoventilation Syndrome; Sleep Apnea, Obstructive; Pulmonary Disease, Chronic Obstructive; Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Full face/Nasal masks (Experimental): Simplus/Eson
  Interventions: Device: Simplus/Eson

INTERVENTIONS:
Device: Simplus/Eson — Released product Simplus and Eson masks

SUMMARY:
This investigation is designed to evaluate the performance, comfort and ease of use of the Simplus and Eson masks amongst NIV patients who are currently on Bi-level therapy

DETAILED DESCRIPTION:
Up to 40 NIV patients who currently use a full face mask or a nasal mask will be recruited. They will be issued a Simplus (if they are existing full face users) or Eson (if they are existing nasal users) to use in-home for 2 weeks. This will consists of male and female participants who have been prescribed with NIV therapy for at least 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18+
* Existing full face mask user or a nasal mask user
* Prescribed NIV therapy for at least 3 months

Exclusion Criteria:

* Inability to give informed consent
* Pregnant or think they may be pregnant
* Anatomical or physiological conditions making NIVtherapy inappropriate
* Patients who are in a coma or decreased level of consciousness
* Existing Simplus and Eson users

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-04; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Objective Leak data | 2 weeks
  Obtained from the participant's device

SECONDARY OUTCOMES:
Subjective measurement of Leak | 2 weeks
  Questionnaire
Subjective measurement of Comfort | 2 weeks
  Questionnaire
Subjective measurement of Ease of Use | 2 weeks
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ingo Fietze, Professor, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No